CLINICAL TRIAL: NCT01216137
Title: The Effects of Vestibular Rehabilitation on MS-related Fatigue and Upright Postural Control: a Randomized Controlled Trial
Brief Title: Effects of Vestibular Rehabilitation on MS-related Fatigue: a Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-1108; PP1501 (Other Grant/Funding Number: National Multiple Sclerosis Society Pilot Research Award)
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Multiple Sclerosis; Fatigue; Balance; Dizziness
Keywords: Multiple Sclerosis; Fatigue; Balance; Upright Postural Control; Dizziness
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Dizziness | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exercise: Vestibular Rehabilitation (Experimental): Balance and eye movement training
  Interventions: Other: Exercise: Vestibular Rehabilitation
- Exercise Control (Active Comparator): Bicycle ergometry and stretching
  Interventions: Other: Exercise
- Wait-listed Control (No Intervention): Wait-listed Control

INTERVENTIONS:
Other: Exercise: Vestibular Rehabilitation — Balance and eye movement training
  Arms: Exercise: Vestibular Rehabilitation
Other: Exercise — Bicycle ergometry and stretching
  Arms: Exercise Control

SUMMARY:
The purpose of this study was to test the feasibility and effectiveness of a novel exercise intervention for individuals who live with multiple sclerosis (MS).

DETAILED DESCRIPTION:
The investigators investigated the effect of a vestibular exercise program designed to help people with MS with two common problems: fatigue and difficulties with balance while standing and walking. Our primary aim was to compare the results from persons with MS that participated in the vestibular exercises (Experimental group) to individuals who participated in a more typical rehabilitation exercise program consisting of stretching and endurance exercise (Exercise Control group) or people who did not receive exercise treatment (Control group).

The study was a 14-week randomized controlled trial. Thirty eighty participants were followed for four weeks before being randomly assigned to one of the three groups. Each participant had an equal chance of being assigned to either the Experimental group, Exercise Control group or the Control group. The Experimental group received a standardized vestibular exercise program that included upright postural control (balance) and eye movement exercises (6 one-hour sessions over 6 weeks). The Exercise Control group received endurance training using a stationary bicycle and leg stretching exercises (6 one-hour sessions over 6 weeks). Both exercise groups received the same 5 minutes of fatigue management education. Measurements of self-reported fatigue, dizziness and depression, and performance of a computerized, standing upright postural control test and walking capacity test were measured to determine benefits from the interventions. Participants in the Control group did not exercise, however if they chose, received the treatment within the clinical setting upon completion of their participation in the study.

The investigators hypothesized that: 1) participants in the Experimental group would improve significantly in fatigue and balance; 2) improvements found in the Experimental group would be significantly greater than improvements in the Exercise Control group and Control group.

Results: Analyses occur at: Baseline; at 10 weeks of follow-up (Baseline to post-intervention; and at 14 weeks of follow-up (post-intervention to post-four week unsupervised follow-up.

ELIGIBILITY:
Inclusion Criteria:

* (1) Clinically definite MS confirmed by a board certified Neurologist
* (2) Kurtzke Expanded Disability Status Scale (EDSS) 0.0 to 6.0 (ranges and corresponding ambulatory status: 0.0 to 4.5 fully ambulatory without assistive device; 5.0 to 5.5 impaired ambulatory status without assistive device; 6.0 impaired ambulatory status with intermittent or unilateral constant assistive device)
* (3) Age: 18 to 65 years (65 years has been set as the upper limit of age to decrease the possible age-related changes in physical strength, endurance, and upright postural control)
* (4) Male or Female (MS affects both gender types)
* (5) Comprehension of the general concept of the study and ability to make informed consent (see Section I. Special Consent Issues). (6) Minorities included
* (7) Self-reported fatigue level on the Modified Fatigue Impact Scale (MFIS) of a total score > 45 (This criterion has been used in previous studies investigating treatment for MS-related fatigue utilizing the MFIS)
* (8) Sensory organization test (SOT) composite score of < 72

Exclusion Criteria:

* (1) Non-ambulatory
* (2) Utilization of agents to control fatigue: i.e. medications: Amantadine, Pemoline, Dexedrine Amphetamine, Methylphenidate, Provigil, Ritalin, Prokarin.
* (3) Utilization of medication(s) that have known possible side effects of fatigue such as: skeletal muscle relaxants (i.e. Baclofen, Zanaflex), Statin Drugs, pain medication (i.e. Opioids, tricyclic antidepressants (TCAs), anti-epileptic drugs (AEDs)
* (4) Any other possible cause of fatigue: major sleep disorder, clinically diagnosed major depressive disorder, anemia, hypothyroidism, B12 deficiency, cancer
* (5) Other neurological disorder which might contribute to significant balance problems, including cerebral vascular accident, peripheral neuropathy (separate from MS diagnosis, such as diabetes mellitus), peripheral vestibular disorders (unilateral/bilateral vestibular hypofunction: benign positional paroxysmal vertigo, Meniere's disease, acoustic neuroma)
* (6) Change in MS specific medication (for disease modification) in the last three months
* (7) Documented MS-related exacerbation in the last six months
* (8) Any medical diagnosis or condition that is considered to be an absolute or relative contraindication to participating in exercise testing and/or result in limitations for participation in an active exercise program or aerobic exercise program, as recommended by the American College of Sports Medicine (ACSM)
* (9) Participation in an exercise routine specifically designed as a vestibular and/or aerobic exercise program within eight weeks prior to study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2007-01; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Self-reported fatigue | 10 weeks
  Modified Fatigue Impact Scale. Analyses occur at: Baseline; at 10 weeks of follow-up (Baseline to post-intervention; and at 14 weeks of follow-up (post-intervention to post-four week unsupervised follow-up.
Upright postural control | 10 weeks
  Sensory Organization Test (SOT)-Posturography. Analyses occur at: Baseline; at 10 weeks of follow-up (Baseline to post-intervention; and at 14 weeks of follow-up (post-intervention to post-four week unsupervised follow-up.
Walking capacity | 10 weeks
  6-minute walk test (6MWT). Analyses occur at: Baseline; at 10 weeks of follow-up (Baseline to post-intervention; and at 14 weeks of follow-up (post-intervention to post-four week unsupervised follow-up.

SECONDARY OUTCOMES:
Self-reported dizziness | 10 weeks
  Dizziness Handicap Inventory. Analyses occur at: Baseline; at 10 weeks of follow-up (Baseline to post-intervention; and at 14 weeks of follow-up (post-intervention to post-four week unsupervised follow-up.
Self-reported depression | 10 weeks
  Beck Depression Inventory - II. Analyses occur at: Baseline; at 10 weeks of follow-up (Baseline to post-intervention; and at 14 weeks of follow-up (post-intervention to post-four week unsupervised follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Schenkman, PT, PhD, Principal Investigator — University of Colorado, Denver

REFERENCES:
- [Derived] Hebert JR, Corboy JR, Manago MM, Schenkman M. Effects of vestibular rehabilitation on multiple sclerosis-related fatigue and upright postural control: a randomized controlled trial. Phys Ther. 2011 Aug;91(8):1166-83. doi: 10.2522/ptj.20100399. Epub 2011 Jun 16. PMID 21680771